CLINICAL TRIAL: NCT00947700
Title: UW ACE Project II, Early Detection and Intervention in Infants at Risk for Autism
Brief Title: Early Connections, Early Detection and Intervention in Infants at Risk for Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); Autism Speaks (Other); Washington State Department of Social and Health Services (Other); Autism Science Foundation (Other)
Responsible Party: Principal Investigator, Sara Jane Webb, Associate Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 32400; P50HD055782 (NIH); P30ES007033 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Infants; Risk markers; ERP; Parent child interaction; Promoting First Relations; Social Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Communication | interventions — Restraint, Physical; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment & Monitoring (No Intervention): No Intervention. Parent-Child participants in assessment and monitoring visits but does not receive any study provided treatment.
- Assessment, Monitoring + Intervention (Experimental): Parent-Child participants in assessment and monitoring visits but also the Promoting First Relationships PFR intervention (http://pfrprogram. Org). PFR is a 10 weekly 60-85 minute in-home visits by a masters level mental health provider trained in the PFR curriculum. The PFR curriculum focuses on increasing parenting sensitivity using attachment theory-informed, strength-based consultation strategies. The curriculum is fully manualized and fidelity was assessed according to the manual.
  Interventions: Behavioral: Assessment, Monitoring & Intervention

INTERVENTIONS:
Behavioral: Assessment, Monitoring & Intervention — Assessment and monitoring at 6, 12, 18 and 24 months; Parent delivered intervention provided between 6 and 12 months.
  Other Names: Promoting First Relationships
  Arms: Assessment, Monitoring + Intervention

SUMMARY:
Early connections has two broad goals:

* to identify risk indices for autism spectrum disorder (ASD) in 6 to 24 month old infants who have an older sibling with ASD or infants who have an older neurotypical sibling.
* to assess whether it is possible to alter risk processes through early intervention with high-risk infants, thereby reducing social-communication delays or the severity of autism symptoms.

DETAILED DESCRIPTION:
Researchers at the University of Washington want to learn more about the benefits of early monitoring and intervention for younger siblings of children with autism spectrum disorders (ASD). The information gained in this study may improve methods of early detection and intervention for infants who may be at risk for developing autism and lead to better outcome for these young children and their families.

Participants include families with a child who has been diagnosed with an autism spectrum disorder or typical development and a younger sibling 12 months old or younger. The study protocol includes: (1) comprehensive infant evaluations at the University of Washington Autism Center at 6-months, 12-months, 18-months and 24-months of age. (2) Developmental screening for the older sibling. (3) Questionnaires and phone interviews for parents. (4) Random assignment to an assessment and monitoring intervention group or a University of Washington intervention group. All families will receive advice regarding appropriate intervention services. Families who are assigned to the UW intervention will take part in a parent delivered intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older sibling with ASD (biologically related to participant)
* Participant 12 months of age or younger
* Within 1 hour of University of Washington
* Interested in participating in Intervention

Exclusion Criteria:

* Out of study area
* Serious parent substance abuse or psychiatric history
* Diagnosis of known genetic syndromes or neurological conditions (infant participant or older sibling)
* Serious motor impairment (infant participant)
* Significant prematurity (infant participant)

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Autism Symptoms | 12 months
  AOSI
Mullen Receptive Language Scale | 12 months
  Mullen Receptive Language Scale SS
Communication and Symbolic Behavior Scale | 12 months
  CSBS Total Composite Score

SECONDARY OUTCOMES:
Parent Child Interaction | 12 months
  NCAST Caregiver Total
Parent quality of life | 12 months
  Questionnaire on Resources and Stress Total Score

CONTACTS AND LOCATIONS:
Overall Officials: Bryan King, MD, Principal Investigator — University of Washington; Sara J Webb, PhD, Principal Investigator — University of Washington; Annette Estes, PhD, Principal Investigator — University of Washington
Locations (1):
- Center on Human Development and Disabilities, University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Participant level data was submitted to NDAR.